CLINICAL TRIAL: NCT05467111
Title: Cardioprotective Effect of Acute Exercise in Breast Cancer Patients
Acronym: CardioProtEx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, Alejandro San Juan Ferrer, PhD Physical Activity and Health, Technical University of Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DATOS-20220624-ASJF-Efecto car
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Early-stage Breast Cancer
Keywords: Breast Cancer; Exercise; Doxorubicin; anthracyclines; Cardiotoxicity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Cardiotoxicity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Patients will perform an acute bout of exercise (different types of exercise for each cycle of anthracyclines) 24-48 hours prior to each cycle of anthracyclines.
  Interventions: Other: Acute Exercise
- Control (No Intervention): Patients will receive standard treatment for each type of tumor proposed by the hospital. This group of patients will be provided with the international recommendations on physical exercise for cancer patients.

INTERVENTIONS:
Other: Acute Exercise — Patients will perform an acute bout of exercise (different types of exercise for each cycle of anthracyclines, as aerobic exercise, strength training or combined training) 24-48 hours prior to each cycle of anthracyclines.
  Arms: Exercise

SUMMARY:
Cardiotoxicity is one of the most significant adverse effects in breast cancer patients treated with anthracyclines (a type of chemotherapy), so we propose to determine whether acute training (i.e., 24h before each chemotherapy session) could reduce the levels of a cardiac biomarker which measures muscle damage (NT-proBNP).

Given the fact NT-proBNP attenuation has been observed with one session performed 24h before the first treatment, we propose to verify these findings in each cycle of doxorubicin analyzing how each type of exercise (aerobic, strength or combined aerobic + strength) may impact on anthracycline-induced cardiotoxicity, since this observation may be relevant considering the feasibility and low cost this implementation would represent in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Woman with non-metastatic breast cancer not previously treated.
* Scheduled to receive neoadjuvant doxorubicin chemotherapy.
* Receive the oncologist´s approval for the practice of exercise.
* Acceptance of randomization.
* To sign an informed consent form before starting any measurement or procedure related to the project.

Exclusion Criteria:

* Patients who receive initial surgery and who are not going to receive neoadjuvant treatment.
* Contraindications to perform stress tests following the recommendations of the American Thoracic Society.
* Pre-existing cardiovascular disease.
* Body mass index (BMI) > 35 kg/m2.
* Diabetes mellitus.
* Renal disease.
* Severe anemia.
* Pregnacy.
* Current smoking status.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
NT-proBNP | 24-48 hours prior to each cycle of anthracyclines and immediately prior to receiving the treatment
  Biomarker of cardiac injury value in blood tests

SECONDARY OUTCOMES:
Cardiac Troponin I | 24-48 hours prior to each cycle of anthracyclines and immediately prior to receiving the treatment
  Biomarker of cardiac injury value in blood tests
Blood Pressure | 24-48 hours prior to each cycle of anthracyclines and immediately prior to receiving the treatment
  Resting blood pressure assesed by sphyngomanometer
Left Ventricular Ejection Fraction (LVEF) | 0-14 days prior to the first treatment ( according to the usual clinical practice) and in the follow-up period (6 months after completion of the anthracycline treatment).
  Change in left ventricular systolic function quantified by transthoracic echocardiography

OTHER OUTCOMES:
Changes in Quality of Life | Prior to each exercise session and in the follow-up period (6 months after completion of the anthracycline treatment).
  Assesed using the validated EORTC-QLQ-C30 quality of life questionnaire
Fatigue | Prior to each exercise session and in the follow-up period (6 months after completion of the anthracycline treatment).
  Assesed using the validated Functional Assessment of Cancer Therapy: Fatigue (FACT-F)
Physical Activity | Prior to each exercise session and in the follow-up period (6 months after completion of the anthracycline treatment).
  Assesed using the validated International Physical Activity Questionnaire (IPAQ-SF)
Assessment of functional mobility | 0-14 days prior to the first treatment and immediately after completion of the anthracycline treatment.
  Assesed using the Timed Up and Go (TUG) test
Assessment of lower extremity strength and power | 0-14 days prior to the first treatment and immediately after completion of the anthracycline treatment.
  Assesed using the Sit to Stand test
Assessment of isometric handgrip | 0-14 days prior to the first treatment and immediately after completion of the anthracycline treatment.
  Assesed using the hand grip dynamometer test

CONTACTS AND LOCATIONS:
Locations (1):
- "Ramón y Cajal" Hospital, Madrid, Spain